CLINICAL TRIAL: NCT04894604
Title: A Prospective, Open, Non-comparative, Post-Market Clinical Follow-up Investigation to Confirm the Safety and Performance of Avance® Solo NPWT System in Surgically Closed Incisions
Brief Title: A Safety and Performance PMCF Investigation of the Avance® Solo NPWT System in Surgically Closed Incisions
Acronym: ASOLO-SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Molnlycke Health Care AB (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-598653
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Incision, Surgical; Surgical Incision; Surgical Wound; Surgical Wound, Recent; Surgical Wound Dehiscence
Keywords: Negative Pressure Wound Therapy; Post Market Clinical Follow-up; Vacuum Assisted Closure
MeSH Terms: conditions — Surgical Wound; Surgical Wound Dehiscence

STUDY DESIGN:
Intervention Model Description: Single group of Subjects (with a low to moderate exuding surgically closed incision) in use of the Avance® Solo NPWT System.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with a low to moderate exuding surgically closed incision (Experimental): Up to 34 study Subjects with a low to moderate exuding surgically closed incision deemed adequate by the Principal Investigator and clinical team for NPWT treatment.
  Interventions: Device: Avance® Solo NPWT System

INTERVENTIONS:
Device: Avance® Solo NPWT System — Application of the Avance® Solo NPWT System on up to 34 study Subjects, in accordance with the IfU for up to 14 days.

SUMMARY:
The ASOLO-SCI investigation is a Post Market Clinical Follow-up (PMCF) study to investigate the safety and performance of the Avance® Solo NPWT System in treating low to moderate exuding surgically closed incisions for up to 14 days when used in accordance with the Instructions for Use (IfU).

DETAILED DESCRIPTION:
The ASOLO-SCI investigation is designed as a prospective, open, non-comparative, PMCF study to investigate the safety and performance of the Avance® Solo NPWT System in treating low to moderate exuding surgically closed incisions for up to 14 days when used in accordance with the IfU in up to 34 patients (n=34).

The ASOLO-SCI investigation is a multicentre study that is expected to take place in approximately three European centres.

The study treatment shall be stopped earlier (i.e. prior to 14 days), in the event study Subjects withdraw their consent, or shall the Principal Investigator and clinical team deem the Avance® Solo NPWT System to be no longer adequate for the study Subject's wound. Following termination of Subject participation for whichever reason in the study, the patient shall be followed in accordance with the local standard of care in wound management and treatment.

As a primary endpoint, the Principal Investigator and clinical team will evaluate whether the surgical incision remains closed, from baseline to study end at Day 14.

ELIGIBILITY:
Inclusion criteria:

1. Male or female ≥ 18 years of age.
2. Signed written Informed Consent Form.
3. Low to moderate exuding surgically closed incisions suitable for suNPWT, according with the Investigator´s judgement and the Avance® Solo NPWT System Instructions for Use.
4. Study subjects that are deemed capable and willing to comply with the protocol instructions.

Exclusion criteria:

1. Known malignancy in the wound or margins of the wound.
2. Untreated and previously confirmed osteomyelitis.
3. Non-enteric and unexplored fistulas.
4. Necrotic tissue with eschar present.
5. Exposed nerves, arteries, veins or organs.
6. Exposed anastomotic site.
7. Known allergy/hypersensitivity to the dressing or its components.
8. Known pregnancy or planning to become pregnant or breastfeeding at time of study participation.
9. Participation in another investigative drug or device trial currently or within the last 30 days.
10. Subjects not suitable for the investigation according to the Investigator's judgement, Clinical Investigation Plan and Instructions for Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in wound remaining closed | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  The evaluation of the wound remaining closed is captured through an assessment by the Principal Investigator/clinical team from baseline to the final visit (wound remaining closed yes/no).

SECONDARY OUTCOMES:
Wound progress to baseline | Day 14 (+0/-2 days)
  Wound progress in low to moderate surgically closed incisions compared between baseline and final visit (deteriorated/no change/improved).
Change in wound progress across visits | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Wound progress in low to moderate surgically closed incisions compared to last visit (deteriorated/no change/improved).
Change in lack of dermal opposition | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Lack of dermal opposition as a percentage of the total wound length from baseline to all follow-up visits.
Change in exudate amount | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Change in exudate amount from baseline to all follow-up visits (none/low/moderate/high).
Change in exudate nature | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Change in exudate nature from baseline to all follow-up visits (serous/fibrinous/serosanguinous/sanguineous/seropurulent/purulent/foul purulent//haemopurulent/haemorrhagic).
Change in exudate odour | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Change in exudate odour from baseline to all follow-up visits (no odour/slight/moderate/strong/very strong).
Change in peri-wound conditions | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Change in peri-wound skin condition from baseline to all follow-up visits (normal/erythematous/oedematous/eczematous/excoriated/macerated/indurated).
Pain assessment | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Subject evaluation of pain at Avance® Solo Border Dressing and Avance® Solo Fixation Strips removal using a Numeric Rating Scale at each follow-up visit (where the Subject verbally grade their pain on a level from 0 to 10, where 0 indicates no pain and 10 the worst imaginable for the Subject; the NRS will be used before and during dressing removal).
Absorption and transportation of exudate | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Clinical assessment of Avance® Solo NPWT System's ability to absorb and/or transport exudate using a rating scale at all follow-up visits (very poor/poor/good/very good).
Trauma to the wound's surrounding skin | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Proportion of Subjects with trauma (e.g. blistering) to the wound site and surrounding skin for Avance® Solo Border Dressing and Avance® Solo Fixation Strips at all follow-up visits.
System wear time | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Evaluate system wear time in days from baseline to all follow-up visits including potential extra visits.
Sounding of alarms | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Subject evaluation of the system properties (number of sounding alarms) assessed at all follow-up visits (souding of alarms in the following intervals 0, 1-5, 6-10, 11-15, 16-20, more than 20).
Product consumption | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Product consumption of the utilised products for the system, from baseline to final visit using the Avance® Solo NPWT System (in total number of Avance® Solo Pumps, Border Dressing, Canisters, Fixation Strips, and batteries).
Subject quality of life assessment | Day 14 (+0/-2 days)
  Subject evaluation of the Avance® Solo NPWT system impact of everyday life at day 14 or final visit. Quality of life is assessed using Numeric Rating Scale (NRS) where the Subject grades how much the treatment has affected their daily life. 0 is equal to no influence, and 10 is equal to considerable influence on everyday life or unbearable. If replying >0, the Subject shall state the presence or absence of the following causes: leakage of dressing, impaired mobility, difficulties in getting dressed, pain, and odour.
Ease of application and removal of the Avance® Solo NPWT System | Baseline, Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Clinician evaluation of ease of application and removal of the Avance® Solo NPWT System using a Numeric Rating Scale collected at baseline and each follow-up visit (from 0 to 10, wherein 0 is equal to no problem with application or removal, and 10 is the worst imaginable situation when applying/removing the system from a Subject).
Subject compliance | Day 7 (+0/-2 days), Day 14 (+0/-2 days)
  Evaluate the Subject compliance to Avance® Solo NPWT System therapy at all follow-up visits by the average number of hours per day that the system has not provided NPWT since the Subject's last visit.
Global satisfaction | Day 14 (+0/-2 days)
  Evaluation of the Principal Investigator and Subject's global satisfactions with the system at day 14 or final visit (very dissatisfied/dissatisfied/neither dissatisfied or satisfied/satisfied/very satisfied).

IPD SHARING:
Plan to Share IPD: No